CLINICAL TRIAL: NCT02870595
Title: The Use of Micro Vibratory Stimulation Technique to Control the Pain of Digit Block Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Christus Spohn Memorial Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 14-007
Record Dates: First submitted 2016-08-11; First posted 2016-08-17 (Estimated); Last update posted 2016-08-17 (Estimated); Status verified 2016-08

CONDITIONS: Pain, Analgesia
MeSH Terms: conditions — Pain; Agnosia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Parallel lidocaine injection (Active Comparator): Informed consent will be obtained from patients undergoing finger local anesthesia digit blocks. Subjects will be randomly assigned (using GraphPAD Randomization Software Tool) to receive the first of their two digit block injections with either the traditional technique (control) or while using the DVICS/ Microvibratory Stimulator. All injections will utilize a 27-gauge needle. The subjects will be given a standard dose of 2mls of 1% lidocaine without epinephrine delivered over 30 seconds. Injections will be timed and performed by a single clinician to avoid large variations in technique and expertise.
  Interventions: Device: Microvibratory Stimulator; Device: Microvibratory Stimulator'
- Parallel (Sham Comparator): In the sham comparator, the device will be placed on the skin, but not turned on. Digit block anesthesia will progress in usual fashion as with active comparator, except without the vibratory device engaged.
  Interventions: Device: Microvibratory Stimulator; Device: Microvibratory Stimulator'

INTERVENTIONS:
Device: Microvibratory Stimulator — Informed consent will be obtained from patients undergoing finger local anesthesia digit blocks. Subjects will be randomly assigned (using GraphPAD Randomization Software Tool) to receive the first of their two digit block injections with either the traditional technique (control) or while using the DVICS/ Microvibratory Stimulator. All injections will utilize a 27-gauge needle. The subjects will be given a standard dose of 2mls of 1% lidocaine without epinephrine delivered over 30 seconds. Injections will be timed and performed by a single clinician to avoid large variations in technique and expertise.
Device: Microvibratory Stimulator' — As above, Microvibratory Stimulator will be used as a sham device in parallel group.

SUMMARY:
The investigators hypothesize that patients who receive 1% lidocaine injections for digit blocks of the finger will experience less pain when the injection is accompanied by the use of a micro-vibratory stimulator (MVS) compared with patients who receive injections without the MVS.

DETAILED DESCRIPTION:
Research Question/Hypothesis

The investigators hypothesize that patients who receive 1% lidocaine injections for digit blocks of the finger will experience less pain when the injection is accompanied by the use of a micro-vibratory stimulator (MVS) compared with patients who receive injections without the MVS.

Objectives

The primary objective of this study is to compare the pain rating scale from an exposure group (digit block injection with the aid MVS) and the control group (traditional injection).

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals between the ages of 18 and 65 who are willing and able to consent and who require the use of local anesthetic digit block to both sides of a finger for the treatment of wounds, injuries, infections, or laceration of the fingers.

Exclusion Criteria:

* Allergy to any type of local anesthetic.
* Inability to Consent.
* Inability to complete a numeric pain scale.
* Clinical appearance or clinical evidence of intoxication.
* Significant compromising conditions such as major trauma and severe respiratory distress.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2014-06; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Pain associated with injection of lidocaine | 30 seconds
  Subjects will rate pain of injection using a 0-10 VAS

IPD SHARING:
Plan to Share IPD: Yes
Data to be published